CLINICAL TRIAL: NCT00691223
Title: Pathogenesis of Focal Dermal Hypoplasia or Goltz Syndrome and Related Disorders
Brief Title: Study of Selected X-linked Disorders: Goltz Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ignatia Van den Veyver, Professor, Baylor College of Medicine
Other Study IDs: BCM Goltz H21291
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Focal Dermal Hypoplasia (FDH); Goltz Syndrome
Keywords: Focal dermal hypoplasia; Goltz syndrome; X linked disorders; PORCN; Wnt signaling
MeSH Terms: conditions — Focal Dermal Hypoplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lymphoblast DNA; tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Individuals with Goltz syndrome and their first degree relatives.

SUMMARY:
Focal dermal hypoplasia, or Goltz syndrome, results from genetic changes, or mutations in the PORCN gene located on the X chromosome. This neurodevelopmental disorder is characterized by birth defects of the skin, skeleton, eyes, and in some cases other organs. Our team is working to obtain a better understanding of how mutations in PORCN lead to the clinical features of Goltz syndrome. We are also trying to identify the genetic change in those patients where no mutations in PORCN have been found. We are also investigating conditions with phenotypes similar to Goltz syndrome to determine if they also have mutations in PORCN. We are collecting blood samples from patients and their parents. DNA from these samples is isolated and then used for genetic testing. We also review medical records to compare clinical symptoms with the detected mutations to determine if there is a correlation.

DETAILED DESCRIPTION:
Goltz syndrome or Focal Dermal Hypoplasia (FDH) is an X-linked dominant neurodevelopmental disorder. The primary features of FDH include areas of hypoplastic skin (atrophy, linear pigmentation and herniation of fat through dermal defects), digital patterning defects (syndactyly, polydactyly, camptodactyly, absence deformities), ocular and dental malformations, mild dysmorphism. Variable other defects include a pointed chin, hypoplastic ears, nasal deformities, short stature, papillomas of lips, gingival and larynx, dystrophic nails, sparse brittle hair. Mental retardation occurs in approximately 15%. 90% of individuals with FDH are female. 95% percent of all cases and 100% of male cases appear de novo.

Using array-based comparative hybridization (array-CGH) a deletion was initially identified in PORCN in two girls with FDH. Sequencing of genes in this region has resulted in the identification of mutations in PORCN in >75% of other individuals affected with FDH. A manuscript describing these mutations was published in Nature Genetics (Wang, 2007). PORCN encodes the human homolog of the Drosophila porcupine protein and has been found in drosophila and mouse studies to be a key regulator of Wnt-protein signaling. We believe that the PORCN mutation may cause FDH by affecting Wnt signaling, but this has yet to be proven.

For this study we are collecting information on patients with clinical findings suggestive of FDH or with known PORCN mutations. A detailed family history will be obtained when indicated, and additional family members will be evaluated afer appropriately obtained written voluntary consent. A detailed report of the history or physical findings will be obtained from referring physicians for patients identified at outside facilities or the participants may be evaluated by the study collaborators. Blood will be obtained from affected individuals unaffected parents and from other affected or unaffected family members where indicated. Occasionally, affected individuals may undergo surgical procedures with removal of tissues; in this case we may obtain tissues that would be otherwise discarded or that are not essential for further diagnostic studies or clinical care of the patient. It is anticipated that these specimens will be extremely valuable for understanding the pathogenesis of the investigated conditions. DNA, RNA or protein will be prepared from leukocytes and from tissues and used for mutation analysis and other molecular studies of the identified genes. Permanent lymphoblastoid cell lines will be prepared and stored in the laboratory as a permanent source of DNA for the molecular studies.

We are not actively recruiting but study remains open for data analysis on existing data and samples.

ELIGIBILITY:
Inclusion Criteria:

* Features suggestive of Goltz syndrome (not all features must be present)

  * Areas of hypoplastic skin
  * Digital patterning defects
  * Ocular and dental malformations
* Presence of a mutation in PORCN

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with Goltz syndrome and their parents. Sometimes additional family members are also enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Identifying the change in the genetic information that causes Goltz syndrome. | Through study completion - average 20 years (recruitment has currently ended)
  The investigators isolate genetic material from samples of individuals with Goltz syndrome and their parents (if available). DNA sequencing and other molecular methods along with bioinformatic analysis is used to find genetic variants (changes) in the genetic code unique to individuals with Goltz syndrome, not seen in healthy population. When a gene that shows variants that are deleterious to its function is identified in at least 3 unrelated Goltz syndrome individuals but not in healthy people (whose DNA sequence is in public databases), the outcome (finding the genetic cause of Goltz syndrome) will be achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Ignatia B Van den Veyver, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified patient data may be published following peer review in journals and/or presented at scientific meetings. There is currently no new recruitment or immediate publication plan.

REFERENCES:
- [Background] Goltz RW. Focal dermal hypoplasia syndrome. An update. Arch Dermatol. 1992 Aug;128(8):1108-11. No abstract available. PMID 1497368
- [Background] GOLTZ RW, PETERSON WC, GORLIN RJ, RAVITS HG. Focal dermal hypoplasia. Arch Dermatol. 1962 Dec;86:708-17. doi: 10.1001/archderm.1962.01590120006002. No abstract available. PMID 13948891
- [Result] Wang X, Reid Sutton V, Omar Peraza-Llanes J, Yu Z, Rosetta R, Kou YC, Eble TN, Patel A, Thaller C, Fang P, Van den Veyver IB. Mutations in X-linked PORCN, a putative regulator of Wnt signaling, cause focal dermal hypoplasia. Nat Genet. 2007 Jul;39(7):836-8. doi: 10.1038/ng2057. Epub 2007 Jun 3. PMID 17546030
- [Result] Ross J, Busch J, Mintz E, Ng D, Stanley A, Brafman D, Sutton VR, Van den Veyver I, Willert K. A rare human syndrome provides genetic evidence that WNT signaling is required for reprogramming of fibroblasts to induced pluripotent stem cells. Cell Rep. 2014 Dec 11;9(5):1770-1780. doi: 10.1016/j.celrep.2014.10.049. Epub 2014 Nov 20. PMID 25464842